CLINICAL TRIAL: NCT04368858
Title: Towards the Use of Instrumented Tests for Screening the Risk of Falling in Patients With Chronic Illness.
Acronym: DETECACTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RBHP 2020 REYNAUD; 2020-A00290-39 (Other: 2020-A00290-39)
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Joint Osteoarthritis; Atherosclerosis of the Distal Arteries, Without Gangrene; Parkinson Disease; Chronic Obstructive Pulmonary Disease, Unspecified; Obesity, Unspecified
Keywords: Inertial sensors; Timed Up and Go test; 6-Minute Walk test; Fall; Risk of fall; Altered mobility; Chronic illness; Chronic pathologies; Physical capacities; Physical test; Activity limitations
MeSH Terms: conditions — Parkinson Disease; Pulmonary Disease, Chronic Obstructive; Obesity; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort 1 : experimental group (Experimental): Participants will be involved in an evaluation program combining, body composition measures, physical tests as well as self-administered questionnaires. Participants will be followed for 1 year with evaluations (occurrence of fall) taking place at 6 months and at 1 year.
  Interventions: Diagnostic Test: Exploratory physiopathology study, including non-invasive functional explorations carried out in patients with chronic pathology.

INTERVENTIONS:
Diagnostic Test: Exploratory physiopathology study, including non-invasive functional explorations carried out in patients with chronic pathology. — In the Mobility Exploration Unit of the University Hospital of Clermont-Ferrand, patients with chronic illnesses undergo a complete assessment of their physical capacities as well as their nutritional status. For the purpose of this protocol, patients will have to perform 2 functional tests, namely the TM6 and the TUG, while being equipped with inertial sensor units (mTUG® and mGAIT®). The data of the gait analysis, posturography and strength analyses as well as the questionnaires' scores will be taken into account in this research. At 6 months and at 1 year, occurrence of a fall will be recorded in order to prospectively monitor this parameter.

SUMMARY:
In patients with chronic illness, screening for falls and their health consequences are major public health issues. Muscle weakness, gait and balance disorders are among the most common risk factors for falling. Assessing these parameters would thus be a crucial step in the evaluation of the risk of falling, allowing to more precisely orient the management strategy. Combining inertial unit sensors with clinically validated tests can provide additional information to improve the assessment of fall risks. We therefore propose to constitute a monocentric exploratory study, testing a prognostic screening tool, in patients suffering from a chronic pathology, in order to assess the risk of falling in this population.

Considering the relationship between muscle weakness and the risk of falling, we can assume that a deficit in muscle strength will result in less vertical acceleration which could point to a muscle cause of the balance disorder and thus allow a finer detection of the risk of falling. On the other hand, we hypothesize that spinal static disorders in chronic pathologies and in particular osteoarthritis, as well as balance disorders linked to impaired deep sensitivity lead to an increase in oscillations of the trunk when walking which can cause postural balance disorders thus increasing the risk of falling.

DETAILED DESCRIPTION:
Investigators propose to constitute a prospective cohort of subjects carrying chronic disease. The main objective is to study the correlation between the vertical acceleration during the sit to stand phase of the instrumented Timed Up and Go test (TUG) and the isokinetic muscle strength of the quadriceps. In addition, as secondary objectives, we will study the potential correlations between the other parameters collected with the inertial sensors during instrumented tests (Timed-Up and Go test, and 6-Minute Walk Test) and the isokinetic muscle strength of the lower limb muscles, posturography parameters, gait parameters, apprehension of fall and others.

In the present protocol, parameters will be measured once at inclusion day (to). Only the falling incidences will be collected prospectively at 6 months and at 1 year from the inclusion day.

Statistical analyses will be carried out using Stata software (version 13, StataCorp, College Station, USA). Qualitative variables will be described in terms of numbers and associated percentages. The quantitative variables will be described in terms of numbers, associated mean and standard deviation, median and interquartile range. Wherever is possible, graphic representations will be associated with these analyses. All tests will be performed for a bilateral hypothesis and a p-value <5% will be considered statistically significant. For the main outcome, the Pearson correlation coefficient (or Spearman if data are not normally distributed) will be calculated with its 95% confidence interval. The analysis of the relationships between the continuous criteria will be carried out using Pearson correlation coefficients (or Spearman if data are not normally distributed).

The search for fall risk factors (at 6 months / 1 year) will be carried out using standard tests:

* Chi-square test (or exact Fisher test when appropriate) for the categorical criteria.
* Student test (or Mann and Whitney test if data not normally distributed) for continuous criteria.

These analyses will be completed using a logistic regression model by adjusting to the clinically relevant criteria or highlighted in the univariate analysis. Results will be presented as an odd ratio with their 95% confidence interval

Little or no missing data is expected on the main criteria, however if a rate of missing data> 5% is observed, a sensitivity analysis for missing data will be carried out in order to characterize their nature (MCAR, MAR, MNAR) in order to propose the most suitable imputation method.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 18 to 90.
* Patients with chronic pathology contributing to impaired mobility.
* Volunteers who have given their written consent.
* Affiliated to French health care system (for France)

Exclusion Criteria:

* Patients suffering from progressive psychiatric pathologies (active psychosis, hallucinations, etc.) or the presence of another serious unstabilized pathology (decompensated heart failure, progressive terminal cancer, etc.).
* People with poorly controlled or unstable cardiovascular disease.
* Major osteoarticular or neurological problems completely preventing the proper performance of the various tests.
* Persons under guardianship, curatorship, deprived of liberty or safeguarding justice.
* People refusing to participate.
* Pregnant or lactating women.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
Vertical acceleration in m/s² during the sit to stand phase of the Timed-Up and Go test. | Day 0
  Vertical acceleration will be collected with the mTUG® inertial sensor unit.
Maximum voluntary isokinetic strength (Nm) of the quadriceps muscles in slow speed (60°/s) concentric contraction. | Day 0
  : Maximum voluntary isokinetic strength of the quadriceps muscles will be measured with the HUMA® /NORM™ device.

SECONDARY OUTCOMES:
Demographics information | day 0
  Demographics information will be obtained using a single questionnaire including questions on age, gender, qualification, personal work status, ethnicity, life and occupational events.
Weight (Kg). | day 0
  Weight will be measured with the medical body weight scale SECA® and according to the ISAK recommendations.
Height (cm). | day 0
  Height will be measured with a wall mounted tape measure and according to the ISAK recommendations.
Waist circumference (cm). | day 0
  Waist circumference will be measured with a medical body tape measure and according to the ISAK recommendations.
Hip circumference (cm). | day 0
  Hip circumference will be measured with a medical body tape measure and according to the ISAK recommendations.
Brachial circumference (cm). | day 0
  Brachial circumference will be measured with a medical body tape measure and according to the ISAK recommendations.
Calf circumference (cm). | day 0
  Calf circumference will be measured with a medical body tape measure and according to the ISAK recommendations.
Body Mass Index (Kg/m²). | day 0
  Description: BMI will be calculated (weight in kilograms divided by height in meters squared).
Body composition. | day 0
  Body composition (muscle and fat) will be measured using he Bodystat® Impedance-meter.
Self-Reported Number of Falls during the previous year | day 0
  Number of falls will be evaluated with the Elderly Fall Screening Test (EFST).
Self-Reported Number of Falls during the previous year | Month 6
  Number of falls will be evaluated with the Elderly Fall Screening Test (EFST).
Self-Reported Number of Falls during the previous year | Year 1
  Number of falls will be evaluated with the Elderly Fall Screening Test (EFST).
Sarcopenia risk. | Day 0
  Sarcopenia risk will be evaluated with the SARC-F Questionnaire.
Balance confidence in performing various activities | Day 0
  Self-report balance confidence will be evaluated with the Activities-specific Balance Confidence (ABC) Scale.
Maximum voluntary isometric strength of the quadriceps muscles at 45° (Nm). | Day 0
  : Maximum voluntary isometric strength of the quadriceps muscles will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the quadriceps muscles at 60°/s (Nm). | Day 0
  Maximum voluntary isokinetic strength of the quadriceps muscles at 60°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the quadriceps muscles at 240°/s (Nm). | Day 0
  Maximum voluntary isokinetic strength of the quadriceps muscles at 240°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the quadriceps muscles at 30°/s (eccentric contraction) (Nm). | Day 0
  Maximum voluntary isokinetic strength of the quadriceps muscles at 30°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the hamstring muscles at 60°/s (Nm). | Day 0
  Maximum voluntary isokinetic strength of the hamstring muscles at 60°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the hamstring muscles at 240°/s (Nm). | Day 0
  Maximum voluntary isokinetic strength of the hamstring muscles at 240°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the hamstring muscles at 30°/s (eccentric contraction) (Nm). | Day 0
  Maximum voluntary isokinetic strength of the hamstring muscles at 30°/s will be measured with the HUMA® /NORM™ device.
Statokinesigram surface area (mm²). | Day 0
  Statokinesigram surface area will be measured with the STATIPRO® static posturography platform.
Stabilogram length (mm). | Day 0
  Stabilogram length will be measured with the STATIPRO® static posturography platform.
Maximal deflection (forward, backward left and right). | Day 0
  Maximal deflection will be measured with the STATIPRO® static posturography platform.
Velocity variations (mm/s). | Day 0
  Velocity variations will be measured with the STATIPRO® static posturography platform.
Romberg ratio according to sway area | day 0
  Romberg ratio will be measured with the STATIPRO® static posturography platform
Romberg ratio according to center of pressure path length. | day 0
  Romberg ratio will be measured with the STATIPRO® static posturography platform.
Plantar pressure ratio sway area. | day 0
  : Plantar pressure ratio sway area will be measured with the STATIPRO® static posturography platform
Plantar pressure ratio length | day 0
  Plantar pressure ratio length will be measured with the STATIPRO® static posturography platform.
Walking velocity (cm/s). | day 0
  Walking velocity will be measured with the GAITRite® Electronic Walkway.
Cadence (steps/min). | day 0
  Cadence will be measured with the GAITRite® Electronic Walkway.
Step length (left and right foot) (cm) | day 0
  : Step length will be measured with the GAITRite® Electronic Walkway.
Stride length (cm). | day 0
  Stride length will be measured with the GAITRite® Electronic Walkway.
: Single support time left and right foot (% of walking cycle) | day 0
  Single support time will be measured with the GAITRite® Electronic Walkway.
Double support time (% of walking cycle). | day 0
  Double support time will be measured with the GAITRite® Electronic Walkway.
Swing time (% of walking cycle). | day 0
  : Swing time will be measured with the GAITRite® Electronic Walkway.
Swing phase (% of walking cycle). | day 0
  Swing phase will be measured with the GAITRite® Electronic Walkway.
Stance phase (% of walking cycle). | day 0
  : Stance phase will be measured with the GAITRite® Electronic Walkway.
Functional capacity Timed-Up and Go | day 0
  Functional capacity will be evaluated using the Timed-Up and Go test.
Functional capacity TDM6 | day 0
  Functional capacity will be evaluated using the 6-minute walk test.
Vertical acceleration (m/s²) during the sit to stand phase of the Timed-Up and Go test (TUG). | day 0
  Vertical acceleration will be measured with the mTUG® inertial sensor unit.
Time (s) to complete the Timed-Up and Go test. | day 0
  Time will be measured with the mTUG® inertial sensor unit.
Anteroposterior acceleration (m/s2) during stand to walk phase of the Timed-Up and Go test | day 0
  Anteroposterior acceleration will be measured with the mTUG® inertial sensor unit.
Vertical angular speed (m/s) during the TUG test. | day 0
  Vertical angular speed will be measured with the mTUG® inertial sensor unit.
Medio-lateral angular velocity (m/s) during the TUG test. | day 0
  Medio-lateral angular velocity (m/s) will be measured with the mTUG® inertial sensor unit.
Time (s) of the 180° rotation phase during the TUG test. | day 0
  Time of the rotation phase will be measured with the mTUG® inertial sensor unit
Time (s) to pass from the sitting position to the first step during the TUG test. | day 0
  Time will be measured with the mTUG® inertial sensor unit.
Duration (s) of the turn to sit phase during the TUG test. | day 0
  Time will be measured with the mTUG® inertial sensor unit.
Total number of steps during the TUG test. | day 0
  Steps will be measured with the mTUG® inertial sensor unit.
Average length of steps (m) during the TUG test. | day 0
  Steps will be measured with the mTUG® inertial sensor unit.
Average walking speed (m/s) during the TUG test. | day 0
  Walking speed will be measured with the mTUG® inertial sensor unit.
Number of steps during the 180° rotation phase of the TUG test. | day 0
  Steps will be measured with the mTUG® inertial sensor unit.
Standard deviation of the duration of the step (s) during the TUG test. | day 0
  Standard deviation will be measured with the mTUG® inertial sensor unit.
Spatio-temporal gait parameters (Average walking speed, step and stride length (right and left), cadence variability, variability in stride length, stance and swing phase, …) during the 6-minute Walk Test (6MWT). | day 0
  Spatio-temporal gait parameters will be measured with the mGAIT® inertial unit sensors

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel COUDEYRE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France